CLINICAL TRIAL: NCT06330350
Title: Investigating Perspectives of Patients With Genodermatosis and Healthcare Professionals on Reproductive Counselling
Brief Title: Qualitative Study in Patients With Genodermatoses and Healthcare Professionals on Reproductive Counselling
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2023-0193
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Quality of Life; Ichthyosis; Palmoplantar Keratoses; Epidermolysis Bullosa; Ectodermal Dysplasia; Basal Cell Nevus Syndrome; Birt-Hogg-Dube Syndrome; Tuberous Sclerosis; Cutis Laxa; Albinism
MeSH Terms: conditions — Ichthyosis; Keratoderma, Palmoplantar; Epidermolysis Bullosa; Ectodermal Dysplasia; Basal Cell Nevus Syndrome; Birt-Hogg-Dube Syndrome; Tuberous Sclerosis; Cutis Laxa; Albinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Keratinisation disorders: Keratinisation disorders comprise a heterogeneous group characterised by abnormal epidermal differentiation, such as variants of ichthyosis and palmoplantar keratoderma.
  Interventions: Other: Qualitative interview
- Skin fragility disorders: Skin fragility disorders comprise a group of inherited blistering diseases, such as variants of epidermolysis bullosa.
  Interventions: Other: Qualitative interview
- Ectodermal dysplasias: Ectodermal dysplasias consists of multiple inherited disorders that are characterised by abnormalities of the embryonic ectoderm, such as hair, nails, sweat glands or teeth.
  Interventions: Other: Qualitative interview
- Dermato-oncogenetic syndromes: This group are genodermatoses associated with the development of malignancies ((non-)cutaneous), such as basal cell nevus syndrome (BCNS), Birt-Hoog-Dubé syndrome, tuberous sclerosis, etc.
  Interventions: Other: Qualitative interview
- Other genodermatoses: In this group genodermatoses are listed that do not fit the other groups as mentioned above, for example albinism and cutis laxa.
  Interventions: Other: Qualitative interview
- Health care professionals: This group includes clinical geneticists, dermatologists and other clinicians involved in the care of patients with genodermatoses.
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Gaining insight into the perspectives of patients with genodermatoses and their partners, and health care professionals concerning reproductive decision-making and counselling.

SUMMARY:
The goal of this observational study is to understand the perspectives and needs of patients with genodermatoses and their partners who wish to have children, regarding their decision-making process and their consideration of reproductive options. Additionally, the investigators aim to investigate the level of knowledge and perspectives of healthcare professionals (such as clinical geneticists, dermatologists and other clinicians involved), and want to explore to what extent patients and their partners are well informed about these reproductive options. To achieve this, the investigators will conduct individual semi-structured qualitative interviews with participants affected by genodermatoses (and their partners) and with healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with genodermatosis (i.e, keratinisation disorders, skin fragility diseases, ectodermal dysplasias, dermato-oncological syndromes, other genodermatoses) and a desire to have children, with if applicable his or her partner with a desire to have children
* Patients with clinically and molecularly confirmed variant of a genodermatosis
* Health care professionals involved with the care of genodermatology patients (e.g. clinical geneticists, dermatologists)

Exclusion Criteria:

* Not being able to communicate verbally in Dutch or English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult patients with genodermatosis (i.e, keratinisation disorders, skin fragility diseases, ectodermal dysplasias, dermato-oncological syndromes, other genodermatoses) and a desire to have children, with if applicable his or her partner with a desire to have children, and health care professionals involved with the care of genodermatology patients (e.g. clinical geneticists, dermatologists).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of perspectives of affected patients + partners and of healthcare professionals concerning reproductive decision-making | 1 day
  Qualitative evaluation of the perspectives and needs of patients with genodermatoses and their partners who wish to have children, as well as clinicians involved in the decision-making process and the consideration of reproductive options, such as prenatal diagnosis (PND), pre-implantation genetic testing (PGT), adoption, the use of donor gametes, refraining from having children, natural pregnancy without genetic testing or foster care. And assessing their level of knowledge on these reproductive options.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gostynski, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands